CLINICAL TRIAL: NCT00123604
Title: Effects of Carvedilol and Metoprolol on Endothelial Function in Hypertensive Patients With Type 2 Diabetes Mellitus
Brief Title: Vascular Effects of Carvedilol Versus Metoprolol in Hypertensive Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Paul Heart Clinic (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Aaron S. Kelly, Ph.D., Senior Research Scientist, St. Paul Heart Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GSK101598
Record Dates: First submitted 2005-07-21; First posted 2005-07-25 (Estimated); Results first posted 2014-11-18 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Hypertension; Type 2 Diabetes Mellitus
Keywords: beta-blockers; endothelial function
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2 | interventions — Carvedilol; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carvedilol (Experimental): Carvedilol, orally, 25 mg, twice daily for five months
  Interventions: Drug: Carvedilol
- Metoprolol (Active Comparator): Metoprolol, orally, 200 mg, twice daily for five months.
  Interventions: Drug: Metoprolol

INTERVENTIONS:
Drug: Carvedilol — 25 mg twice daily for five months.
  Other Names: Coreg
  Arms: Carvedilol
Drug: Metoprolol — 200 mg twice daily for five months.
  Other Names: Lopressor
  Arms: Metoprolol

SUMMARY:
The purpose of this study is to compare the vascular effects of two commonly used blood pressure medications, carvedilol and metoprolol in hypertensive patients with type 2 diabetes.

DETAILED DESCRIPTION:
Carvedilol and metoprolol are two commonly used blood pressure medications that have both been shown to be effective in controlling hypertension. Although in the same drug class, preliminary data have shown that these medications may have different vascular effects. This study will assess which medication is better at improving artery health independent of their blood pressure lowering effects. Artery health will be assessed non-invasively by ultrasound. Certain markers of atherosclerosis found in the blood will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-80 years old
* Documented history of type 2 diabetes
* Stable angiotensin converting enzyme/angiotensin receptor blocker (ACE/ARB) regimen 30 days before and throughout the study period
* Stable anti-diabetic regimen throughout the study period
* Body mass index (BMI) between 22-45 kg/m2
* HbA1c between 6-9% for patients on anti-diabetic treatment regimen and HbA1c between 6-8% for patients who are being controlled by diet alone
* Screening blood pressure (BP) > 130/80 (average of 3 sitting measurements), with current medications

Exclusion Criteria:

* Uncontrollable or symptomatic arrhythmias
* Unstable angina
* Sick sinus syndrome or second or third degree heart block
* Decompensated heart failure
* Myocardial infarction (MI) or stroke within 3 months of screening
* Bradycardia
* Chronic obstructive pulmonary disease (COPD) with required inhaled or oral bronchodilators or corticosteroids
* Bronchial asthma or related bronchospastic conditions
* New onset/diagnosed type 2 diabetes (<3 months)
* Clinically significant renal or liver disease (creatinine >2.5 mg/dL)
* Endocrine disorders
* Use of anorectic or other diet drugs inconsistent with recommendations for type 2 diabetics
* Use of beta-blockers within 3 months of screening
* Use of corticosteroids
* Systemic disease, including cancer, with reduced life expectancy (<12 months)
* Psychological illness/condition that interferes with comprehension of study requirements
* Use of an investigational drug within 30 days of entry into study

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-06; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan J Bank, M.D., Principal Investigator — St. Paul Heart Clinic
Locations (1):
- St. Paul Heart Clinic, Saint Paul, Minnesota, United States

REFERENCES:
- [Derived] Bank AJ, Kelly AS, Thelen AM, Kaiser DR, Gonzalez-Campoy JM. Effects of carvedilol versus metoprolol on endothelial function and oxidative stress in patients with type 2 diabetes mellitus. Am J Hypertens. 2007 Jul;20(7):777-83. doi: 10.1016/j.amjhyper.2007.01.019. PMID 17586413

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occured at medical clinics.
Groups:
- Metoprolol: Metoprolol, orally, 200 mg, once daily
- Carvedilol: Carvedilol, orally, 25 mg, once daily
Period: Overall Study
Arm/Group | Metoprolol | Carvedilol
Started | 19 | 17
Completed | 18 | 16
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Metoprolol: Metoprolol, orally, 200mg, twice daily for five months
- Carvedilol: Carvedilol, orally, 25mg, twice daily for five months
- Total: Total of all reporting groups
Arm/Group | Metoprolol | Carvedilol | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 16 | 34
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (9.9) | 60.9 (8.5) | 61.4 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 13 | 13 | 26
Region of Enrollment [Number; unit: participants]
  United States | 19 | 17 | 36

OUTCOME MEASURES:

1. Primary Outcome: Flow Mediated Dilation
Description: Flow mediated dilation is a measure of endothelial function. It is measured by the percent change in artery diameter (i.e. dilation), pre and post manual artery occlusion.
Time Frame: change from baseline to 5 months
Measure: Mean (Standard Deviation); unit: percentage of change in dilation
Groups:
- Carvedilol: Carvedilol, orally, 25mg, once daily
- Metoprolol: Metoprolol, orally, 200mg, once daily
Arm/Group | Carvedilol | Metoprolol
Number analyzed (Participants) | 16 | 18
percentage of change in dilation | 6.2 (3.9) | 4.1 (3.4)

ADVERSE EVENTS:
Arm/Group | Metoprolol | Carvedilol
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/17
Other Adverse Events (participants affected / at risk) | 0/19 | 0/17

LIMITATIONS AND CAVEATS:
The sample size was relatively small

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No